CLINICAL TRIAL: NCT02524808
Title: Multicentric Project for the Prospective Identification and Validation of Molecular Alterations That Define the "BRCANess" Profile in Ovarian Epithelial Cancer and Its Application as a Response Predictor to Platinum and Antitarget Therapies in the Clinical Practice. The Finding BRCANess Project
Brief Title: Prospective Identification and Validation of "BRCANess" Profile in Ovarian Epithelial Cancer
Acronym: FindBRCANess
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación de investigación HM (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: ESR-14-10537
Record Dates: First submitted 2015-08-06; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational prospective study. Patients diagnosed with advanced epithelial ovarian cancer (stage IC or higher) since 2008 will be asked to participate in this study by signing an informed consent. Tumour samples will be reviewed to confirm the diagnosis and to select the best regions for tissue sampling to perform the following molecular studies: array-based Comparative Genomic Hybridization and Next Generation Sequencing. Detected mutations will be analysed by Sanger sequencing. FISH probes will be designed and tested on the samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced epithelial ovarian cancer (stage IC or higher).

Exclusion Criteria:

* Non

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with advanced epithelial ovarian cancer (stage 1c or higher) since 2008
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a genetic profile defined by sequencing that could predict Progression Free Survival (PFS) | 1 year
  Clinical data from the enrolled patients will be recorded and related to the results obtained from sequencing the DNA isolated from tumor samples. Whole exome sequencing (WES) will be used for sequencing DNA isolated from paraffin embedded samples and Whole genome association study (GWAS) for the DNA from frozen samples. The bioinformatics analysis of the sequencing results will allow us to identify altered regions and affected genes and the minimal common regions of imbalance. All detected mutations will be confirmed by Sanger sequencing to ensure the reliability of the findings.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario HM Sanchinarro - Clara Campal Comprehensive Cancer Center, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complejo Hospitalario de Navarra, Pamplona